CLINICAL TRIAL: NCT04151134
Title: Evaluation of the Role of Tongue Base MucOsectomy and Step sErial Sectioning in the Management of the Unknown Primary Squamous Cell Cancer in the Head and Neck
Brief Title: Evaluation of Tongue Base MucOsectomy & Step sErial Sectioning
Acronym: MOSES
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Oracle Cancer Trust (Unknown); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5065
Record Dates: First submitted 2019-10-10; First posted 2019-11-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tonsil and tongue base resection specimens,buccal swab and/or blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Step serial sectioning histological processing — Step serial sectioning histological processing

SUMMARY:
Squamous cell carcinoma (SCC) is a cancer that originates from the cells lining the body and can spread into the lymph glands and beyond. Some patients first present with an SCC which has moved to the lymph glands of the neck. Clinical examination and imaging investigations are performed to try and identify the site where the cancer has originated. However, if no original site can be identified, then the investigators call these 'cancers of an unknown primary' (CUP) of the head and neck.

One region where these cancers could have originated from is the oropharynx. There are two areas in the oropharynx were cancers commonly arise. One area is the palatine tonsils, which can be removed for analysis with an operation called tonsillectomy. The other area is the tissue lining the back of the tongue, known as the tongue base. A relatively new surgical technique called 'tongue base mucosectomy' (TBM) allows removal of this tissue to see if the primary cancer is contained within it. This study will then use a histological method called 'step serial sectioning' (SSS) to look in more detail at the tonsils and tongue base, hoping to increase the detection rate of the primary cancer.

Centres performing TBM will be asked to participate. Patients will be asked to consent to their tissue being used for SSS after it has undergone conventional histology. Anonymised samples will be sent to a central laboratory in Newcastle for processing. Other anonymised data regarding the patients' diagnosis and care will be collated. Patients will be asked to complete questionnaires regarding pain and swallowing recovery following surgery. A smaller cohort of patients will also be interviewed as part of a qualitative research process to establish their views on CUP and the acceptability of the above treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 or over
* Both sexes
* Cervical metastatic SCC, confirmed with cytology or biopsy, undergoing TBM for identification of primary site

Exclusion Criteria:

* Primary site identified by any means prior to being indicated for TBM
* Patients undergoing targeted biopsies or resections
* Patients known to have a history of previous H&N cancers
* Patients known to have undergone previous radiation to the H&N region

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cervical metastatic SCC, confirmed with cytology or biopsy, undergoing TBM for identification of primary site
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Primary Cancers Identified | Within one year of surgery
  Cancer identified in tonsil and tongue base resections

SECONDARY OUTCOMES:
Pain after tongue base mucosectomy | week 0 , 3 weeks, 6 weeks, 12 weeks, 26 weeks and 52 weeks
  Numeric Pain Scale. A person rates their pain on a scale of 0 to 10
Swallow function after tongue base mucosectomy | week 0 , 3 weeks, 6 weeks, 12 weeks, 26 weeks and 52 weeks
  Patients will be given the MDADI questionnaire in which they will be asked a series of questions with the following possible answers: completely agree, agree, uncertain, disagree, completely disagree

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT04151134/Prot_001.pdf